CLINICAL TRIAL: NCT00655707
Title: A Phase I/II Safety and Tolerability Dose Escalation Study Following the Autologous Infusion of Expanded Adult Haematopoietic Stem Cells to Patients With Liver Insufficiency
Brief Title: A Phase I/II Safety and Tolerability Dose Escalation Study of Autologous Stem Cells to Patients With Liver Insufficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHSC/001
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Liver Disease
Keywords: Adult stem cell therapy
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous CD34+ cells (Experimental): Autologous Cluster Designation 34+(CD34+) cells
  Interventions: Biological: Autologous Expanded CD34+ Haemopoietic cells

INTERVENTIONS:
Biological: Autologous Expanded CD34+ Haemopoietic cells — Autologous expanded CD34+ cells obtained by leukapheresis on a single occasion by infusion into the hepatic artery or portal vein.
  Patient numbers 01 and 02 will receive 1x109 cells Patient numbers 03 and 04 will receive 1x1010 cells Patient numbers 05 and 06 will receive 2x1010 cells Patient numbers 07 and 08 will receive 5x1010 cells

SUMMARY:
This is a prospective dose escalation study of the administration of adult human stem cells in patients with end stage liver failure. Successive groups of two patients will receive ascending doses of autologous adult human stem cells starting at 1x10[9] cells. Following expansion in an approved Good Manufacturing Practice (GMP) facility the cells will be infused into either the hepatic artery or portal vein of research participants.

The aim of this trial is to determine the maximum tolerated dose of autologous adult stem cells when infused into either the hepatic artery or the portal vein. The maximum dose that would be given would be 5x10 to the ten [10].

To assess improvement in liver function as measured by serological and biochemical analysis and determine whether there are any symptomatic improvements as reported by the patients.

DETAILED DESCRIPTION:
This is a prospective dose escalation study of the administration of expanded autologous adult human stem cells in patients with chronic liver insufficiency. Four groups of two patients will receive ascending doses of autologous adult human stem cells starting at a dose of 1 x 10[8] cells. The cells will be infused into either the hepatic artery or the portal vein of research participants. The consultant radiologist will review a duplex Doppler scan of the blood supply to the liver to determine the safest route for delivery of the cells.

The first patients (01 and 02) will receive 1 x 10[8] cells. If no adverse events are observed in either patient in the two-week period post stem cell administration, patient numbers 03 and 04 will receive 5 x 1[08] cells. This will continue through patients 05 and 06 receiving cells at 1 x 10[9] and 07 and 08 receiving 5 x 10[9] cells. If any patient in any cohort suffers adverse events considered to be treatment-related, the next group of patients will receive cells at a concentration one step down from that received by the patient suffering the adverse events.

At the completion of this first stage of the study, if no adverse treatment related events are seen, a further group of 10 patients will receive cells at a concentration of 5 x 10[9] cells.

It should be noted that if fewer cells are obtained at the end of the expansion period the re-infusion of the cells to the patient should nonetheless continue. This patient will be considered inevaluable and the next participant will be allocated their trial number.

The total period that each patient will be participating in the study is 12 weeks and the total duration of this clinical trial is expected to be approximately 12 months.

All patients will be assessed 4 weeks after coming off study (week 12), whether from completion of protocol or early withdrawal for whatever reason. They will also be monitored in the clinic for the remainder of their life.

Patients who are withdrawn due to issues of toxicity will be followed until the adverse event is resolved or the outcome is known. Patients will then be followed-up for four weeks after resolution and thereafter for life in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged from 20 to 65 years of age
* Evidence of chronic liver insufficiency
* The presence of abnormal serum albumin and/or bilirubin and/or prothrombin time
* Patient is unlikely to receive a liver transplant
* Has a World Health Organisation (WHO) performance score of less than 2
* Has a life expectancy of at least 3 months
* Ability to give written consent
* Women of childbearing potential may be included, but must use a reliable and appropriate contraceptive method

Exclusion Criteria:

* Patients below the age of 20 or above the age of 65 years
* Pregnant or lactating women
* Patients with recent recurrent GI bleeding or spontaneous bacterial peritonitis
* Patients with evidence of HIV or other life threatening infection
* Patients unable to give written consent
* Patients with a history of hypersensitivity to Granulocyte-Colony Stimulating Factor (F-CSF)
* Patients who have been included in any other clinical trial within the previous month

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nagy Habib, ChM FRCS, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The planned dose escalation design did not work due to low participants number. All participants received similar dose of Autologous expanded CD34+ cells .
Groups:
- Treatment: Autologous CD34+ cells
  Autologous Expanded CD34+ Haemopoietic cells: Autologous expanded CD34+ cells obtained by leukapheresis on a single occasion by infusion into the hepatic artery or portal vein.
Period: Overall Study
Arm/Group | Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Autologous CD34+ Cells: Patients enrolled in the study underwent 5 days of treatment with G-CSF to mobilise CD34+ cells, followed by leukapheresis to obtain CD34+ cells.
Arm/Group | Autologous CD34+ Cells
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] — 20 - 65 years patients
  years | 49.4 [42 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Tolerated the Maximum Dose
Description: To determine the maximum tolerated dose of autologous adult stem cells when infused into either the hepatic artery or the portal vein.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Autologous CD34+ Cells: Autologous Expanded CD34+ Haemopoietic cells: Autologous expanded CD34+ cells obtained by leukapheresis on a single occasion by infusion into the hepatic artery or portal vein.
Arm/Group | Autologous CD34+ Cells
Number analyzed (Participants) | 5
Participants | 5

2. Primary Outcome: Number of Participants Without Specific Treatment Related Side Effect
Description: To assess the safety of ascending doses of autologous adult stem cells when introduced into either the hepatic artery or the portal vein and to determine the maximum tolerated dose of stem cells.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Autologous CD34+ cells
  Autologous expanded CD34+ cells obtained by leukapheresis on a single occasion by infusion into the hepatic artery or portal vein.
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Autologous CD34+ Cells
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous CD34+ Cells (N=5)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) — Urinary tract infection requiring hospitalisation and antibiotic administration.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous CD34+ Cells (N=5)
Fever (Immune system disorders) | 4 (4) — Mild fever following stem cell injection
Pain (Surgical and medical procedures) | 4 (4) — Mild abdominal pain reported following the stem cell injection
Nausea (Gastrointestinal disorders) | 5 (5) — Nausea following stem cell injection
Jaundice (Hepatobiliary disorders) | 1 (4) — Mild jaundice occurred following the stem cell injection
Ascites (Hepatobiliary disorders) | 3 (3) — Mild ascvited developed following stem cell injection

LIMITATIONS AND CAVEATS:
This was not a randomised study and although the results were encouraging only a small number of patients were treated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes